CLINICAL TRIAL: NCT04766840
Title: A Study to Evaluate the Safety and Efficacy of Donor-derived CAR-T Cells in the Treatment of Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Donor-derived CAR-T Cells in the Treatment of AML Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YMCART202005
Record Dates: First submitted 2021-01-27; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-01

CONDITIONS: AML
Keywords: CAR-T; Immunotherapy
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM73 CAR-T (Experimental): Drug: IM73 CAR-T Cells
  * Fludarabine
  * Cyclophosphamide
  Interventions: Drug: CAR-T cells

INTERVENTIONS:
Drug: CAR-T cells — Drug: IM73 CAR-T Cells Drug: Fludarabine Two days before cell infusion, patient will be treated with fludarabine for 3 days Drug: Cyclophosphamide: Two days before cell infusion, patient will be treated with Cyclophosphamide for 3 days
  Other Names: IM73 CAR-T Cells

SUMMARY:
This is a clinical study to evaluate the safety and efficacy of donor-derived CAR-T cells in the treatment of patients with relapsed or refractory acute myeloid leukemia in China.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label study. This study is planned to enroll about 9 subjects with relapsed or refractory acute myelogenous leukemia and 9 matched donors for leukapheresis and CAR-T cells manufacture. Donor-derived CAR-T cells were then infused intravenously into subjects, in a dose-escalating 3+3 design.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or relapsed AML patients.
* Have found an appropriate matched donor for CAR-T cells manufacturing.
* Patients must have evaluable evidence of disease.
* Age ≥ 18 years; Expected survival is more than 3 months.
* ECOG score 0-2 points.
* Women of childbearing age have negative blood pregnancy test before the start of the trial, and agree to take effective contraceptive measures during the trial until the last follow-up; male subjects with partners of childbearing potential agree to take effective contraceptive measures during the trial until the last follow-up.
* Adequet liver, kidney, heart and lung function.

Exclusion Criteria:

* Confirmed acute promyelocytic leukemia; or recent symptomatic central nervous system leukemia.
* Patients with graft-versus-host disease requiring the use of immunosuppressive agents; or patients with autoimmune system diseases.
* Prior use of any gene therapy product.
* History of epilepsy or other central nervous system diseases.
* Presence of concurrent active malignancy.
* Active hepatitis B or C virus, patients with HIV or syphilis infection.
* Currently participating in or having participated in other drug clinical trials during past 30 days.
* Active or uncontrolled infection requiring systemic therapy within 14 days prior to enrollment.
* Other situations not suitable for the study judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | 28 days
  ≥ Grade 4 adverse event related to CAR-T cells infusion

SECONDARY OUTCOMES:
Objective response rate | 28 days
  Patients who achieve CR（complete response） or CRi 28 days after CAR-T cells infusuion

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital (PKUPH), Beijing, China

IPD SHARING:
Plan to Share IPD: No